CLINICAL TRIAL: NCT03711903
Title: A Phase 2, Randomized, Double Blind, Placebo , Controlled Study To Evaluate The Administration of CN-105 In Participants With Acute Supratentorial Intracerebral Hemorrhage
Brief Title: Evaluation of CN-105 in Subject With Acute Supratentorial Intracerebral Hemorrhage
Acronym: S-CATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Collaborators: AegisCN LLC (Industry); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: S-CATCH
Record Dates: First submitted 2018-09-28; First posted 2018-10-19 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The treatment arm will be given CN 105 The placebo arm will be give 0/9% NaCl
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): The study drug, CN-105, will be administered at 1.0 mg/kg every 6 +/- 1 hour. The calculated volumes of study agent will be removed from the vials and transferred to 250 mL of normal saline (0.9% sodium chloride injection, USP). The recorded weight at baseline will be used to determine the appropriate amount of CN-105 drug product to administer. Estimated weight may be used if recorded weight is not available. Each dose of CN-105 or placebo will be administered as a slow IV bolus over 30 minutes.
  Interventions: Drug: Acetyl-Valine-Serine-Arginine-Arginine-Arginine-NH2 (Ac-VSRRR- NH2).
- Placebo arm (Placebo Comparator): The Placebo arm will be given 0.9% NaCL
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: Acetyl-Valine-Serine-Arginine-Arginine-Arginine-NH2 (Ac-VSRRR- NH2). — The study drug, CN-105 is supplied in amber glass vials containing 4 mL of a concentrated 12.5-mg/mL clear-to-slightly-yellow solution.
  Other Names: CN105
  Arms: Treatment arm
Drug: 0.9% Sodium-chloride — normal saline
  Arms: Placebo arm

SUMMARY:
Phase 2, randomized, double-blind, placebo controlled study to evaluate the administration of CN-105 in patients with supratentorial intracerebral hemorrhage (ICH). Patients will be evaluated for eligibility within 12 hours of symptom onset. Eligible participants (30 active participants and 30 control participants) will receive CN-105 or placebo administered intravenously (IV) for a 30-minute infusion every 6 hours for up to a maximum of 3 days (13 doses) or until discharge (if earlier than 3 days). Participants will be monitored daily throughout the Treatment phase of the study (up to a maximum of 5 days) and will receive standard-of-care treatment for the duration of the study. Additional protocol assessments will be required during the Treatment phase as outlined in Section 7.5. After discharge from the hospital, participants will enter a 3-month Follow-up phase, with a clinic visit at 30 days and a follow-up telephone interview with telephone-validated mRS at 90 days after first dose of study agent.

DETAILED DESCRIPTION:
Phase 2, randomized, double-blind, placebo controlled study to evaluate the administration of CN-105 in patients with supratentorial intracerebral hemorrhage (ICH). Patients will be evaluated for eligibility within 12 hours of symptom onset. Eligible participants (30 active participants and 30 control participants) will receive CN-105 or placebo administered intravenously (IV) for a 30-minute infusion every 6 hours for up to a maximum of 3 days (13 doses) or until discharge (if earlier than 3 days). Participants will be monitored daily throughout the Treatment phase of the study (up to a maximum of 5 days) and will receive standard-of-care treatment for the duration of the study. Additional protocol assessments will be required during the Treatment phase as outlined in Section 7.5. After discharge from the hospital, participants will enter a 3-month Follow-up phase, with a clinic visit at 30 days and a follow-up telephone interview with telephone-validated mRS at 90 days after first dose of study agent.

The study is not powered to test any specific hypothesis in regard to safety and will instead use descriptive methods to describe the experience of the study cohort with respect to adverse and serious adverse events (SAEs), as well as the occurrence of several pre-specified events of interest. The secondary objective of this study will be met by comparing the modified Rankin score (mRS) at 30 days between participants treated with CN-105 with placebo controlled participants The mRS at 30 days will be compared between treated and control participants using the Wilcoxon rank sum test. Exploratory analyses include comparison of treated and control participants for radiographic cerebral edema and hematoma volume and expansion and biological markers of inflammation.

Primary: To assess safety of CN-105 administration in primary ICH.

Secondary: To evaluate whether the administration of CN-105 improves 30-day mortality and functional outcomes by comparing participants treated with CN-105 with placebo controlled participants.

Exploratory:

* To investigate feasibility of Day 0, 1, 2, and 5 non-contrast head computed tomography (CT) as a radiographic surrogate to evaluate progression of perihematomal edema
* To investigate feasibility of using serial biochemical markers of neuroinflammation and neuronal injury as a surrogate measure of perihematomal edema and clinical outcome in the setting of spontaneous ICH.Primary:
* Number and severity of AEs throughout the duration of the study
* Number and severity of SAEs throughout the duration of the study
* In-hospital, 30-day, and 90-day mortality
* Treatment-related mortality
* In-hospital neurological deterioration, defined as an increase of National Institutes of Health Stroke Scale (NIHSS), > 2 from baseline and/or decrease of > 2 of Glasgow Coma Scale (GCS), persisting more than 24 hours, and unrelated to sedation
* Incidence of cerebritis, meningitis, ventriculitis
* Incidence of systemic infection
* Incidence of hematoma extension Secondary:.
* 30- and 90-day mRS
* Need for intracranial hypertension management
* NIHSS score, Glasgow Coma Scale, Montreal Cognitive Assessment, Stroke Impact Scale-16, and Barthel Index assessment at hospital discharge and 30 days after ICH
* Discharge disposition

Exploratory:

* Day 0, 1, 2, 5 non-contrast head CT as a radiographic surrogate to evaluate progression of perihematomal edema
* Biochemical surrogates of brain injury, including plasma concentrations of S100B, glial fibrillary acidic protein, metalloproteinase-3 and -9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin-6, tumor necrosis factor-α, and vascular endothelial growth factor, assessed daily for 5 days after ICH or until discharge (concentration time area under the curve assessed for each biomarker)

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent to participate in the study in accordance with required regulations; if a participant is not capable of providing informed consent, written consent must be obtained from the participant's legally authorized representative (LAR).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Is male or female, age 30 to 80 years, inclusive.
4. Has a confirmed diagnosis of spontaneous supratentorial ICH.
5. Able to receive first dose of study drug ≤ 12 hours after onset of ICH symptoms, such as alteration in level of consciousness, severe headache, nausea, vomiting, seizure, and/or focal neurological deficits, or last-known well time.
6. Has an interpretable and measurable diagnostic CT scan.
7. Has a GCS score ≥ 5 on presentation
8. Has a National Institutes of Health Stroke Scale (NIHSS) score ≥ 4
9. Has systolic BP (SBP) < 200 mm Hg at enrollment.

Exclusion Criteria:

1Known pregnancy and lactation 2.Has a temperature greater than 38.5°C at Screening. 3.ICH known to result from trauma. 4.Evidence of infratentorial hemorrhage (any involvement of the midbrain or lower brainstem as demonstrated by radiograph or complete third nerve palsy) severely limiting the recovery potential of the patient in the opinion of the investigator.

5.Evidence of primary intraventricular hemorrhage deemed to be at high risk for obstructive hydrocephalus, in the opinion of the investigator or evidence of extra-axial (i.e., subarachnoid or subdural) extension of hemorrhage severely limiting the recovery potential of the patient in the opinion of the investigator.

6.Radiographic evidence of underlying tumor. 7.Known unstable mass or active radiographic evidence and symptoms of herniation syndromes severely limiting the recovery potential of the patient in the opinion of the investigator.

8.Known ruptured aneurysm, arteriovenous malformation, or vascular anomaly. 9.Has a platelet count < 100,000/mL. 10.Has an international normalized ratio (INR) > 1.5 or irreversible coagulopathy either due to medical condition or detected before screening.

11.Is taking new oral anticoagulants (NOACS) or low molecular weight heparin at the time of ICH onset 12.In the opinion of the investigator is unstable and would benefit from supportive care rather than supportive care plus CN-105.

13. In the opinion of the investigator has any contraindication to the planned study assessments, including CT and MRI.

14.Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which, in the opinion of the investigator, unacceptably increases the individual's risk by participating in the study.

15.Concomitant enrollment in another interventional study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
adverse event | 0-12 hours
  any untoward medical occurrence associated with the use of the drug in a participant
adverse event | 24 hour
  untoward medical occurrence associated with the use of the study drug whether considered related or not
adverse event | 48 hour
  untoward medical occurrence associated with the use of the study drug whether considered related or not
adverse event | 72 hour
  untoward medical occurrence associated with the use of the study drug whether considered related or not
adverse event | 96 hour
  untoward medical occurrence associated wtth the use of study drug whether considered related or not
adverse event | 120 hour
  untoward medical occurrence associated wtth the use of study drug whether considered related or not
adverse event | 30 day
  untoward medical occurrence associated with the use of study drug whether considered related or not
adverse event | 90 day
  untoward medical occurrence associated with the use of study drug whether considered related or not
GCS | 0-12 hour
  score as per scale
GCS | 24H
  scored as per scale
GCS | 48 hours
  scored as per scale
GCS | 72 Hour
  scored as per scale
GCS | 96 hour
  scored as per scale
GCS | at 120 hour
  scored as per scale
GCS | at 30 day
  scored as per scale
NIHSS | 0- 12 hour
  scored as per assessment
NIHSS | 120 hour
  scored as per assessment
NIHSS | 24 hour
  scored as per assessment
NIHSS | 48 hour
  scored as per assessment
NIHSS | 72 hour
  scored as per assessment
NIHSS | 96 Hour
  scored as per assessment
NIHSS score | 30 day
  score as per assessment
Serious adverse event | 48 hour
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | 0-12 hour
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | 72 hour
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | 96 hour
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | at 90 day
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | at 120 hour
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
Serious adverse event | at 30 day
  An AE is considered serious if the investigator believes any of the following outcomes may occur: death, life threatening AE which places participants at immediate risk of death at the time of the event as it occurred, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; Congenital abnormality or birth defect ;Requires inpatient hospitalization or prolongation of existing hospitalization with the exception or preplanned (before the study) hospital admissions, planned admissions, hospitalization of less then 24 hours (after discharge from index hospitalization.
systemic infection | 0-12 hour
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 24 hour
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 48 hour
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 72 hour
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 96 hours
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 120 hours
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 30 day
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
systemic infection | 90 day
  presence of any infection supported by clinical diagnosis, or any laboratory work up.
Brain CT scan | 0-12 hour
  evaluate hematoma expansion
Brain CT scan | 24 Hour
  evaluate hematoma expansion
presence of CNS infection | 24 hour
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 72 hours
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 0-12 hour
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 48 hours
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 120 hour
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 96 hour
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 30 day
  meningitis, cerebritis, ventriculitis
presence of CNS infection | 90 day
  meningitis, cerebritis, ventriculitis
Mortality | 0-12 hour
  death related or unrelated to the study drug
Mortality | 48 hour
  death related or unrelated to the study drug
Mortality | 72 hour
  death related or unrelated to the study drug
Mortality | 24 hour
  death related or unrelated to the study drug
Mortality | 96 hour
  death related or unrelated to the study drug
Mortality | 120 hour
  death related or unrelated to the study drug
Mortality | 30- day
  occurrence of death related or not related to the use of the study drug
Mortality | 90 -day
  occurrence of death related or not related to the use of the study drug

SECONDARY OUTCOMES:
outcome as assessed by mRS | 120 hour
  MRS scoring
functional outcome as assessed by mRS | 30 Day
  MRS scoring
outcome as assessed by mRS | 90Day
  MRS scoring
cognitive assessment | 120 Hour
  Montreal cognitive assessment
Discharge disposition | day 90
  The place where the patient was discharge -either home, nursing home or rehabilitation care facilities
cognitive assessment | 30 day
  Montreal cognitive assessment
Barthel index | 120 hour
  score as per assessment
Barthel index | 30 day
  score as per assessment
Barthel index | 90 day
  score as per assessment

OTHER OUTCOMES:
biomarkers of brain injury | 0-12 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor
biomarkers of brain injury | 24 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor
biomarkers of brain injury | 48 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor
biomarkers of brain injury | 72 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor
biomarkers of brain injury | 96 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor
biomarkers of brain injury | 120 hour
  plasma concentrations of s100 B, glial fibrillary acidic protein, metalloproteinase -3 and 9, C-reactive protein, D-dimer, brain natriuretic peptide, interleukin -6, tumor necrosis factor, and vascular epithelial growth factor

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li N, Liu YF, Ma L, Worthmann H, Wang YL, Wang YJ, Gao YP, Raab P, Dengler R, Weissenborn K, Zhao XQ. Association of molecular markers with perihematomal edema and clinical outcome in intracerebral hemorrhage. Stroke. 2013 Mar;44(3):658-63. doi: 10.1161/STROKEAHA.112.673590. Epub 2013 Feb 6. PMID 23391772
- [Background] Lynch JR, Pineda JA, Morgan D, Zhang L, Warner DS, Benveniste H, Laskowitz DT. Apolipoprotein E affects the central nervous system response to injury and the development of cerebral edema. Ann Neurol. 2002 Jan;51(1):113-7. doi: 10.1002/ana.10098. PMID 11782990
- [Background] Lynch JR, Wang H, Mace B, Leinenweber S, Warner DS, Bennett ER, Vitek MP, McKenna S, Laskowitz DT. A novel therapeutic derived from apolipoprotein E reduces brain inflammation and improves outcome after closed head injury. Exp Neurol. 2005 Mar;192(1):109-16. doi: 10.1016/j.expneurol.2004.11.014. PMID 15698624
- [Background] Wang J, Dore S. Inflammation after intracerebral hemorrhage. J Cereb Blood Flow Metab. 2007 May;27(5):894-908. doi: 10.1038/sj.jcbfm.9600403. Epub 2006 Oct 11. PMID 17033693
- [Background] Gao J, Wang H, Sheng H, Lynch JR, Warner DS, Durham L, Vitek MP, Laskowitz DT. A novel apoE-derived therapeutic reduces vasospasm and improves outcome in a murine model of subarachnoid hemorrhage. Neurocrit Care. 2006;4(1):25-31. doi: 10.1385/NCC:4:1:025. PMID 16498192
- [Background] Aono M, Bennett ER, Kim KS, Lynch JR, Myers J, Pearlstein RD, Warner DS, Laskowitz DT. Protective effect of apolipoprotein E-mimetic peptides on N-methyl-D-aspartate excitotoxicity in primary rat neuronal-glial cell cultures. Neuroscience. 2003;116(2):437-45. doi: 10.1016/s0306-4522(02)00709-1. PMID 12559098
- [Background] Gebel JM Jr, Jauch EC, Brott TG, Khoury J, Sauerbeck L, Salisbury S, Spilker J, Tomsick TA, Duldner J, Broderick JP. Relative edema volume is a predictor of outcome in patients with hyperacute spontaneous intracerebral hemorrhage. Stroke. 2002 Nov;33(11):2636-41. doi: 10.1161/01.str.0000035283.34109.ea. PMID 12411654
- [Background] Carhuapoma JR, Barker PB, Hanley DF, Wang P, Beauchamp NJ. Human brain hemorrhage: quantification of perihematoma edema by use of diffusion-weighted MR imaging. AJNR Am J Neuroradiol. 2002 Sep;23(8):1322-6. PMID 12223372
- [Result] Guptill JT, Raja SM, Boakye-Agyeman F, Noveck R, Ramey S, Tu TM, Laskowitz DT. Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety, Tolerability, and Pharmacokinetics of a Single Escalating Dose and Repeated Doses of CN-105 in Healthy Adult Subjects. J Clin Pharmacol. 2017 Jun;57(6):770-776. doi: 10.1002/jcph.853. Epub 2016 Dec 19. PMID 27990643
- [Result] Laskowitz DT, Goel S, Bennett ER, Matthew WD. Apolipoprotein E suppresses glial cell secretion of TNF alpha. J Neuroimmunol. 1997 Jun;76(1-2):70-4. doi: 10.1016/s0165-5728(97)00021-0. PMID 9184634
- [Result] Lei B, James ML, Liu J, Zhou G, Venkatraman TN, Lascola CD, Acheson SK, Dubois LG, Laskowitz DT, Wang H. Neuroprotective pentapeptide CN-105 improves functional and histological outcomes in a murine model of intracerebral hemorrhage. Sci Rep. 2016 Oct 7;6:34834. doi: 10.1038/srep34834. PMID 27713572
- [Result] Misra UK, Adlakha CL, Gawdi G, McMillian MK, Pizzo SV, Laskowitz DT. Apolipoprotein E and mimetic peptide initiate a calcium-dependent signaling response in macrophages. J Leukoc Biol. 2001 Oct;70(4):677-83. PMID 11590206
- [Result] Laskowitz DT, Wang H, Chen T, Lubkin DT, Cantillana V, Tu TM, Kernagis D, Zhou G, Macy G, Kolls BJ, Dawson HN. Neuroprotective pentapeptide CN-105 is associated with reduced sterile inflammation and improved functional outcomes in a traumatic brain injury murine model. Sci Rep. 2017 Apr 21;7:46461. doi: 10.1038/srep46461. PMID 28429734
- [Result] Laskowitz DT, Thekdi AD, Thekdi SD, Han SK, Myers JK, Pizzo SV, Bennett ER. Downregulation of microglial activation by apolipoprotein E and apoE-mimetic peptides. Exp Neurol. 2001 Jan;167(1):74-85. doi: 10.1006/exnr.2001.7541. PMID 11161595
- [Result] Laskowitz DT, Blessing R, Floyd J, White WD, Lynch JR. Panel of biomarkers predicts stroke. Ann N Y Acad Sci. 2005 Aug;1053:30. doi: 10.1196/annals.1344.051. No abstract available. PMID 16179504
- [Result] Lynch JR, Blessing R, White WD, Grocott HP, Newman MF, Laskowitz DT. Novel diagnostic test for acute stroke. Stroke. 2004 Jan;35(1):57-63. doi: 10.1161/01.STR.0000105927.62344.4C. Epub 2003 Dec 11. PMID 14671250